CLINICAL TRIAL: NCT03843671
Title: A Phase II Randomized Sham-Controlled Trial With Allocation Concealment and Blinded Patients and Assessors, Investigating Hyperbaric Oxygen as a Radiation Sensitizer for Locally Advanced Squamous Cell Carcinoma of the Oropharynx and Larynx
Brief Title: Hyperbaric Radiation Sensitization of Head and Neck Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Baromedical Services (Other)
Collaborators: Mayo Clinic (Other); Dartmouth-Hitchcock Medical Center (Other); CISSS de Chaudière-Appalaches (Other Government); Memorial Hermann Hospital (Other); David Grant U.S. Air Force Medical Center (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency); Prisma Health Richland Hospital (Unknown); William Jennings Bryan Dorn VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NBS2019-1; 93840508 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2019-02-04; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Hyperbaric oxygen; HNSCC; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized sham-controlled, with allocation concealment and blinded patients and assessors
Who Masked: Participant, Outcomes Assessor
Masking Description: Both groups compressed in a hyperbaric chamber. Patients will be unaware of the compression gas or degree of pressurization as references to each are obscured
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Experimental): Hyperbaric oxygen Hyperbaric chamber
  Interventions: Drug: Hyperbaric oxygen; Device: Hyperbaric chamber
- Group 2 (Sham Comparator): Sham for hyperbaric oxygen Hyperbaric chamber
  Interventions: Drug: Hyperbaric oxygen; Device: Hyperbaric chamber

INTERVENTIONS:
Drug: Hyperbaric oxygen — Hyperbaric oxygen therapy
  Other Names: Hyperbaric chamber
Device: Hyperbaric chamber — Hyperbaric chamber

SUMMARY:
There is reason to believe that hyperbaric oxygen administered immediately prior to radiotherapy will prove beneficial for this cancer type and stage. The basis for this hypothesis is a review of several decades of published work, the conclusion of a recent (2018) Cochrane Review, and results of a Phase I trial.

DETAILED DESCRIPTION:
The goal of this research is to address the question:

"Does the addition of hyperbaric oxygen to radiation and chemotherapy improve outcomes in locally advanced oropharyngeal or laryngeal squamous cell carcinoma?"

There is reason to believe that hyperbaric oxygen administered immediately prior to radiotherapy will prove beneficial for this cancer type and stage. The basis for this hypothesis is a review of several decades of published work, the conclusion of a recent (2018) Cochrane Review, and results of a Phase I trial. A summary of this body of work follows.

During the 1950's, several reports laid the groundwork for hyperbaric oxygen's potential as an effective radiation sensitizer. Gray and colleagues observed that curability of small animal tumors with radiotherapy was limited by the radio-resistance of the portion of cells that retain their reproductive integrity.(1) Tumor cell sensitivity to irradiation was seen to increase when tumor-bearing mice breathed oxygen under hyperbaric conditions. Gray's group further observed that radiobiological damage demonstrates dependence on the concentration of oxygen in the immediate vicinity of tumor cells at the time of radiation.( 2) It became evident that many solid tumor cell populations exist within a wide range of oxygen tensions.(3) These findings were sufficiently encouraging to warrant a small clinical study to determine if this anticipated radio-sensitization effect could be demonstrated histologically.(4) A small diver recompression chamber was acquired from the Royal Navy and modified to accommodate a recessed acrylic window.(5)

The trial involved eight patients whose breast or lung tumor sites would lie directly below the window, above which a radiation delivery source was mounted. To assess any difference afforded by hyperbaric oxygen, tumors had to be large enough so they could addressed in two aspects. Irradiation of the inferior aspect occurred conventionally, with the superior aspect shielded. Shielding was then reversed and the superior aspect irradiated while patients breathed oxygen to 3.0 atmospheres absolute.(4) Preliminary findings of increased tumor destruction secondary to hyperbaric oxygen exposure promoted investigators to treat another 35 patients in this manner. Despite their uniformly poor prognosis, the hyperbaric effect was again significant and outcomes were deemed "much better than anticipated".(6)

On the strength of this preliminary data there was widespread interest in hyperbaric radiation sensitization.(7,8,9,10) However, frustration at the lack of 'visibility' for other anatomic sites with these chamber types initially limited wider application. Industry responded by manufacturing purpose-built chambers with increasing numbers of windows. By the early 1960's, a completely seamless acrylic hyperbaric chamber had been produced.

It eventually became apparent that hyperbaric oxygen's effectiveness was inconsistent across all tumor types (the concept of varying tumor hypoxic fraction was in its infancy). Quite probably, many of these cancers had already metastasized. Along with suggestions of a higher incidence of new primary tumors and rates of metastasis in hyperbaric oxygen irradiated patients, (11, 12) the testing of alternative sensitizers, and a lack of uniformity in radiation dosing (making comparisons difficult), interest in hyperbaric sensitization eventually began to wane. By the early 1970's, the hyperbaric chamber as a sensitizing agent had largely been abandoned.

Little more was heard of this sensitization technique until 1996, when Japanese neurosurgeons reported the results a small clinical trial investigating malignant gliomas.(13) Due to the evolution of targeted radiation delivery devices it was no longer possible to undertake concurrent hyperbaric oxygen and radiotherapy. This group, therefore, introduced a sequential approach, irradiating patients immediately upon exiting the chamber. They were encouraged enough by their findings to undertake, along with several other Japanese groups, additional brain tumor trials.

In 1997, Machin et al. summarized 30 years of the U.K.'s Medical Research Council sponsored trials of solid tumors, using modern statistical methodology.(14) When the five trials involving hyperbaric sensitization were re-analyzed, a clear survival advantage was evident in each of the two head and neck cancer trials, with mixed results in cancers of the cervix. In 1999, oncologists from Yale reported the results of a head and neck squamous cell carcinoma trial, conducted 20 years earlier.(15) Patients were randomized to receive radiotherapy conventionally or during hyperbaric oxygenation. Significant improvement in local control, and relapse free survival at five years was evident in the hyperbaric group.

In 2000, magnetic resonance imaging demonstrated hyperbaric oxygen's ability to elevate implanted tumor oxygen levels in mice. This effect remained for 20-30 minutes after chamber decompression.(16) Malignant glioma oxygen responses to various conditions were measured via stereotactic CT guided implanted oxygen electrodes in 18 patients.(17) Hyperbaric, but not normobaric, oxygen significantly increased tumor oxygen tension, and this effect likewise remained for more than 20 minutes following patient removal from the chamber. This study had involved pre- and post-hyperbaric recordings. Becker and colleagues took this one step further and measured tumor oxygen response prior to and during hyperbaric oxygen exposure.(18) In seven head and neck squamous cell carcinoma patients, mean baseline tumor oxygen pressure was 17 mmHg, increasing to 550 mmHg in a mean of 17 minutes of hyperbaric oxygen breathing.

Four clinical trials have further evaluated the sensitization potential of hyperbaric oxygen in malignant gliomas. This technique was considered feasible, held promise,(19) and involved minimal toxicity,(20,21) and modestly extended overall survival.(19,20,21,22)

A 2018 Cochrane Review concluded that 'given the findings of improved tumor control and mortality with the use of hyperbaric oxygen for patients with cancers of the head and neck…, there is a case for large randomized trials of high methodological vigor…'.(23)

In contrast to earlier unsystematic reports, a 2003 meta-analysis failed to establish a causal relationship between hyperbaric oxygen therapy and de novo development of a tumor, established tumor growth, or an increase in the degree of metastases.(24)

Key messages from this body of work:

i. Radiation-resistance is largely a function of tumor tissue hypoxia ii. Hyperbaric oxygen elevates squamous cell carcinoma oxygen tension in animals and man.

iii. In humans, squamous cell carcinoma oxygen tensions to peak at a mean of 17 minutes during hyperbaric oxygenation. They remain elevated for more than 15 minutes after exposure.

iv. Provision of hyperbaric oxygen has proven feasible and safe as a radiation sensitizer for both malignant brain tumors and head and neck squamous cell carcinomas.

In preparation for this Phase II trial, a Phase I 'dose escalation' study was undertaken.(25) Its purpose was to verify safety and tolerability of hyperbaric oxygen immediately prior to radiation therapy for oropharyngeal carcinoma. It also assessed the acute toxicity impact of hyperbaric oxygen delivered in different groups twice, three times, and five times weekly. With a mean follow-up of 19 months, five days per week hyperbaric dosing had not increased overall toxicity, and patient compliance was good. (25) Complete clinical response occurred in all patients who completed the protocol. One patient suffered bone and liver metastases. While this study was not designed to assess clinical outcomes, a subsequent report involving a minimum 61 months follow-up confirmed no late toxicities, with overall survival of 100%, zero local recurrence, and an 11% incidence of distant metastases.(26)

Citations are listed in the Reference section

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological or microscopic proof (from the primary tumor and/or lymph nodes) of invasive squamous cell carcinoma of the oral cavity, oropharynx or larynx (World Health Organization type 1).
2. Stage III or IV disease, M0
3. Non-surgical candidate; for reasons of health or age (except biopsy)
4. Human Papillomavirus (P16) negative
5. Life expectancy of at least 6 months and a Karnofsky performance status of ≥ 70
6. Age ≥ 18 years
7. No distant metastatic disease
8. No clinically significant heart disease:

   No significant ventricular arrhythmia requiring medication with antiarrhythmic. No symptomatic coronary artery disease (angina). No myocardial infarction within the last 6 months. No second or third degree heart block or bundle branch block or clinically significant conduction system abnormality.
9. Patients must sign a study-specific informed consent form

Exclusion Criteria:

1. Histology other than squamous cell carcinoma
2. Evidence of metastasis (below the clavicle or distant) by clinical or radiographic means
3. History of prior invasive malignancy, unless at least 5 years without evidence of recurrence (tumor-specific restaging)
4. Prior resection of the primary tumor or lymph node, unless un-operated N2-N3 nodal disease or primary tumor remaining, respectively.
5. Prior chemotherapy for head and neck cancer or radiotherapy to the head and neck
6. Prior treatment with Bleomycin
7. Creatinine clearance: measured or estimated Glomerular Filtration Rate <40 ml/min.
8. Patients with simultaneous primaries
9. Pregnancy
10. Participating in a conflicting protocol
11. Pulmonary pathologies (risk of decompression-induced pulmonary barotrauma)

    Current, untreated pneumothorax. Previous history of spontaneous pneumothorax. Previous history of intrathoracic surgery. History or evidence of pulmonary blebs or bullous lung disease. Clinically significant chronic obstructive pulmonary disease, associated with carbon dioxide retention, poorly controlled or associated with acute bronchospasm.
12. Where the hyperbaric physician deems the patient to have an otherwise unacceptable risk for hyperbaric chamber exposure
13. Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Two years
  Per blinded radiotherapy assessor
Relapse free survival | Two years
  Per blinded radiotherapy assessor

SECONDARY OUTCOMES:
Overall survival | Two years
  Per blinded radiotherapy assessor
Incidence of acute hyperbaric complications; ear/sinus barotrauma, oxygen toxicity, myopia, confinement anxiety | At seven weeks from start of protocol, having completed 35 hyperbaric chamber exposures
  Clinical and study record assessment by hyperbaric physician
Incidence and degree of acute radiation toxicity | At seven weeks from start of protocol, having completed 35 radiotherapy treatments
  Common Terminology Criteria Adverse Events version 5.0
Incidence and degree of late radiation tissue injury | Two years
  Common Terminology Criteria Adverse Events version 5.0 and clinical assessment
Hyperbaric protocol and radiotherapy dosing protocol compliance | Approximately 45 days after initiation of protocol
  Assessed per Radiation Therapy Chair and hyperbaric oxygen physician per medical record review
Subject quality of life: Rating scale | Two week post RT, then 3, 6, 12 & 24 months post radiotherapy
  Functional Assessment of Cancer Therapy: Head and Neck version 4.0 $ Performance Status Scale for Head and Neck.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Clarke, Study Chair — National Baromedical Services; James R Hussey, PhD, Principal Investigator — University of South Carolina School of Public Health; James Wells, MD, Principal Investigator — Dorn Veterans Medical Center; Lindsie Cone, MD, Principal Investigator — Prisma Health Richland Hospital
Locations (5):
- United States (4):
  - The Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Wilford Hall Medical Facility, San Antonio, Texas
- Hotel Dieu Hospital of Levis, Lévis, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GRAY LH. Radiobiologic basis of oxygen as a modifying factor in radiation therapy. Am J Roentgenol Radium Ther Nucl Med. 1961 May;85:803-15. No abstract available. PMID 13708070
- [Background] GRAY LH, CONGER AD, EBERT M, HORNSEY S, SCOTT OC. The concentration of oxygen dissolved in tissues at the time of irradiation as a factor in radiotherapy. Br J Radiol. 1953 Dec;26(312):638-48. doi: 10.1259/0007-1285-26-312-638. No abstract available. PMID 13106296
- [Background] GRAY LH. Oxygenation in radiotherapy. I. Radiobiological considerations. Br J Radiol. 1957 Aug;30(356):403-6. doi: 10.1259/0007-1285-30-356-403. No abstract available. PMID 13446401
- [Background] CHURCHILL-DAVIDSON I, SANGER C, THOMLINSON RH. High-pressure oxygen and radiotherapy. Lancet. 1955 May 28;268(6874):1091-5. doi: 10.1016/s0140-6736(55)90589-4. No abstract available. PMID 14382503
- [Background] CHURCHILL-DAVIDSON I, SANGER C, THOMLINSON RH. Oxygenation in radiotherapy. II. Clinical application. Br J Radiol. 1957 Aug;30(356):406-22. doi: 10.1259/0007-1285-30-356-406. No abstract available. PMID 13446402
- [Background] EMERY EW, LUCAS BG, WILLIAMS KG. Technique of irradiation of conscious patients under increased oxygen pressure. Lancet. 1960 Jan 30;1(7118):248-50. doi: 10.1016/s0140-6736(60)90170-7. No abstract available. PMID 13820164
- [Background] SANGER C. High pressure oxygen and radiation therapy. Am J Roentgenol Radium Ther Nucl Med. 1959 Mar;81(3):498-503. No abstract available. PMID 13627317
- [Background] ATKINS HL, SEAMAN WB, JACOX HW, MATTEO RS. EXPERIENCE WITH HYPERBARIC OXYGENATION IN CLINICAL RADIOTHERAPY. Am J Roentgenol Radium Ther Nucl Med. 1965 Mar;93:651-63. No abstract available. PMID 14258312
- [Background] CATER DB, SCHOENIGER EL, WATKINSON DA. Effects on oxygen tension of tumours of breathing oxygen at high pressures. Lancet. 1962 Aug 25;2(7252):381-3. doi: 10.1016/s0140-6736(62)90233-7. No abstract available. PMID 13877337
- [Background] Evans JC. Metastasis following radiotherapy in hyperbaric oxygen. Radiology. 1969 Nov;93(5):1155-7. doi: 10.1148/93.5.1155. No abstract available. PMID 5350691
- [Background] Johnson RE, Kagan AR, Bryant TL. Hyperbaric oxygen effect on experimental tumor growth. Radiology. 1967 Apr;88(4):775-7. doi: 10.1148/88.4.775. No abstract available. PMID 6020944
- [Background] Kohshi K, Kinoshita Y, Terashima H, Konda N, Yokota A, Soejima T. Radiotherapy after hyperbaric oxygenation for malignant gliomas: a pilot study. J Cancer Res Clin Oncol. 1996;122(11):676-8. doi: 10.1007/BF01209031. PMID 8898978
- [Background] Machin D, Stenning SP, Parmar MK, Fayers PM, Girling DJ, Stephens RJ, Stewart LA, Whaley JB. Thirty years of Medical Research Council randomized trials in solid tumours. Clin Oncol (R Coll Radiol). 1997;9(2):100-14. doi: 10.1016/s0936-6555(05)80448-0. PMID 9135895
- [Background] Haffty BG, Hurley R, Peters LJ. Radiation therapy with hyperbaric oxygen at 4 atmospheres pressure in the management of squamous cell carcinoma of the head and neck: results of a randomized clinical trial. Cancer J Sci Am. 1999 Nov-Dec;5(6):341-7. PMID 10606475
- [Background] Kohshi K, Kinoshita Y, Imada H, Kunugita N, Abe H, Terashima H, Tokui N, Uemura S. Effects of radiotherapy after hyperbaric oxygenation on malignant gliomas. Br J Cancer. 1999 Apr;80(1-2):236-41. doi: 10.1038/sj.bjc.6690345. PMID 10390002
- [Background] Kinoshita Y, Kohshi K, Kunugita N, Tosaki T, Yokota A. Preservation of tumour oxygen after hyperbaric oxygenation monitored by magnetic resonance imaging. Br J Cancer. 2000 Jan;82(1):88-92. doi: 10.1054/bjoc.1999.0882. PMID 10638972
- [Background] Beppu T, Kamada K, Yoshida Y, Arai H, Ogasawara K, Ogawa A. Change of oxygen pressure in glioblastoma tissue under various conditions. J Neurooncol. 2002 May;58(1):47-52. doi: 10.1023/a:1015832726054. PMID 12160140
- [Background] Becker A, Kuhnt T, Liedtke H, Krivokuca A, Bloching M, Dunst J. Oxygenation measurements in head and neck cancers during hyperbaric oxygenation. Strahlenther Onkol. 2002 Feb;178(2):105-8. doi: 10.1007/s00066-002-0892-0. PMID 11942033
- [Background] Ogawa K, Yoshii Y, Inoue O, Toita T, Saito A, Kakinohana Y, Adachi G, Ishikawa Y, Kin S, Murayama S. Prospective trial of radiotherapy after hyperbaric oxygenation with chemotherapy for high-grade gliomas. Radiother Oncol. 2003 Apr;67(1):63-7. doi: 10.1016/s0167-8140(02)00406-1. PMID 12758241
- [Background] Beppu T, Kamada K, Nakamura R, Oikawa H, Takeda M, Fukuda T, Arai H, Ogasawara K, Ogawa A. A phase II study of radiotherapy after hyperbaric oxygenation combined with interferon-beta and nimustine hydrochloride to treat supratentorial malignant gliomas. J Neurooncol. 2003 Jan;61(2):161-70. doi: 10.1023/a:1022169107872. PMID 12622455
- [Background] Ogawa K, Yoshii Y, Inoue O, Toita T, Saito A, Kakinohana Y, Adachi G, Iraha S, Tamaki W, Sugimoto K, Hyodo A, Murayama S. Phase II trial of radiotherapy after hyperbaric oxygenation with chemotherapy for high-grade gliomas. Br J Cancer. 2006 Oct 9;95(7):862-8. doi: 10.1038/sj.bjc.6603342. Epub 2006 Sep 5. PMID 16953239
- [Background] Kohshi K, Yamamoto H, Nakahara A, Katoh T, Takagi M. Fractionated stereotactic radiotherapy using gamma unit after hyperbaric oxygenation on recurrent high-grade gliomas. J Neurooncol. 2007 May;82(3):297-303. doi: 10.1007/s11060-006-9283-1. Epub 2006 Nov 22. PMID 17120158
- [Background] Bennett M, et al. Hyperbaric Oxygenation for Tumor Sensitization to Radiotherapy. In The Cochrane Library, Issue 1, 2006. Oxford: Update Software. 1-61.
- [Background] Feldmeier J, Carl U, Hartmann K, Sminia P. Hyperbaric oxygen: does it promote growth or recurrence of malignancy? Undersea Hyperb Med. 2003 Spring;30(1):1-18. PMID 12841604
- [Background] Hartford AC, Davis TH, Buckey JC, Foote RL, Sinesi MS, Williams BB, Fariss AK, Schaner PE, Claus PL, Okuno SH, Hussey JR, Clarke RE. Hyperbaric Oxygen as Radiation Sensitizer for Locally Advanced Squamous Cell Carcinoma of the Oropharynx: A Phase 1 Dose-Escalation Study. Int J Radiat Oncol Biol Phys. 2017 Mar 1;97(3):481-486. doi: 10.1016/j.ijrobp.2016.10.048. Epub 2016 Nov 15. PMID 28126298